CLINICAL TRIAL: NCT04539652
Title: A Multicenter, Single-Arm, Phase 4 Clinical Trial to Evaluate the Efficacy and Safety of TenofoBell® Tablet in Chronic Hepatitis B Patients in Treatment of Oral Antiviral Therapy for Hepatitis B Virus
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of TenofoBell® Tablet in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 285HBV18018
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Experimental

INTERVENTIONS:
Drug: Experimental — Experimental group are treated with TenofoBell®

SUMMARY:
This study was designed to evaluate the rate of subjects with HBV DNA less than 20 IU/mL after taking TenofoBell® tablet for 48 weeks

ELIGIBILITY:
1. Inclusion Criteria:

1. Patients who show positive HBsAg
2. Patients who show positive or negative HBeAg

2. Exclusion Criteria:

1. Patients who have hepatitis C(HCV), hepatitis D(HDV) or human immunodeficiency virus(HIV)
2. Patients with a history of allergic reaction to Tenofovir
3. Patients who are unable to participate in clinical trials based on investigator's decision.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Rate of subjects with HBV DNA less than 20 IU/mL | change after 48 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Daegu Chatholic University Medical center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No